CLINICAL TRIAL: NCT04648774
Title: Continuous Serratus Anterior Blockade for Sternotomy Analgesia Following Cardiac Surgery: A Pilot Feasibility Study.
Brief Title: Continuous Serratus Anterior Blockade for Sternotomy
Acronym: Cardiac-SAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSH REB#1026626
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Pain; Opioid Use; Quality of Life
Keywords: cardiac surgery; regional anesthesia; fascial plane block; enhanced recovery after surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: A computer-generated random number will be assigned and tracked by the central pharmacy to randomize patients on a 1:1 basis to the Ropivacaine and placebo groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Nova Scotia Health (NSH) pharmacy will prepare either Ropivacaine 0.2% (2mg/ml) or normal saline in identical bags labelled as "study drug" such that the patient, clinical staff and the researchers are blinded to assigned group. The pharmacy will maintain the assignment list, only unmasking assignment in cases of suspected local anesthetic systemic toxicity (LAST) or allergic reactions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active serratus anterior plane (SAP) block with Ropivacaine 0.2% (Active Comparator)
  Interventions: Procedure: Serratus anterior plane (SAP) block
- Placebo serratus anterior plane (SAP) block with normal saline (Placebo Comparator)
  Interventions: Procedure: Normal saline placebo

INTERVENTIONS:
Procedure: Serratus anterior plane (SAP) block — With the patient in supine position, an ultrasound transducer will be used to find the 4th rib in the mid-axillary line. A 17g touhy needle will be introduced in-plane in an inferior to superior direction until its tip rests between the serratus anterior muscle and the 4th rib or the 3rd external intercostal muscle. A bolus of study drug 10ml (either ropivacaine 0.2% or normal saline) will be delivered though the needle. A 18g multiholed catheter will be inserted and secured to the patients' skin with adhesive dressings. A further 10ml of study drug will be administered through the catheter. The same procedure will be followed on the contralateral side. The study drug will be administered by programmed intermittent bolus (PIB) 10ml every 2 hours to each side in a staggered, alternating fashion. The PIB study drug will to be continued for 72 hours post-insertion.
  Arms: Active serratus anterior plane (SAP) block with Ropivacaine 0.2%
Procedure: Normal saline placebo — Patients in both groups will receive the standard of care analgesic medications in the cardiovascular intensive care unit and the ward.
  Arms: Placebo serratus anterior plane (SAP) block with normal saline

SUMMARY:
This is a pilot study to assess the feasibility of a full study. The purpose is to assess the analgesic effectiveness of the serratus anterior plane (SAP) block following cardiac surgery.

Patients will be randomized to receive either Ropivacaine 0.2% or placebo via bilateral SAP block catheters for 72 hours postoperatively.

DETAILED DESCRIPTION:
Inadequate pain relief following cardiac surgery increases morbidity, length of stay in the intensive care unit, persistent pain, and costs. Moderate to severe pain is common after cardiac surgery, peaking during the first and second postoperative day, then decreasing after the third day.

Regional anesthesia as part of a multimodal pain management strategy has become a key feature of cardiac surgery enhanced recovery after surgery (ERAS) protocols. A technique consolidating the pectoralis nerve block (PECS) and serratus anterior plane block (SAPB) into a single injection has been described, also called the serratus anterior plane (SAP) block. Given the relative paucity of evidence assessing the utility of continuous serratus anterior plane block (cSAP) in cardiac surgery, we decided to assess the feasibility of a placebo controlled randomized controlled trial (RCT) with a pilot study.

Primary Pilot Study Objective To assess feasibility of a larger intervention study by measuring recruitment rate, adherence rate, retention rates and continuous serratus anterior plane block (cSAP)-related adverse events following cardiac surgery via median sternotomy.

Methods This study will include patients undergoing valvular replacement/repair and/or coronary artery bypass grafting (CABG) at the QEII Health Sciences Center in Halifax, Nova Scotia. The study will include a maximum of 50 participants, randomly assigned to 2 study arms of 25 participants. A computer-generated random number will be assigned by the central pharmacy to randomize patients on a 1:1 basis to the Ropivacaine and placebo groups.

cSAP block procedure - Study Intervention A member of the cardiac anesthesia or regional anesthesia team will place bilateral serratus anterior catheters under ultrasound guidance within 2 hours of arrival to the cardiovascular intensive care unit. A bolus of study drug 20ml (either ropivacaine 0.2% or normal saline) will be delivered at the time of the block. A 18g multiholed catheter will be inserted and secured to the patients' skin. The same procedure will be followed on the contralateral side. The study drug will be administered by programmed intermittent bolus (PIB) 10ml every 2 hours to each side in a staggered, alternating fashion. The PIB study drug will to be continued for 72 hours post-insertion.

Feasibility endpoints The study will be deemed feasible if it meets the following predetermined endpoints: 1. Recruitment of 4 patients per month; 2. The adherence rate to protocols is >90%; 3. Primary outcome measurement rate is >90%; 4. Combined major catheter-related adverse event rate (pneumothorax + LAST + allergic reaction) is <2%.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged >18 years) patients at time of screening
* Undergoing valvular replacement/repair and/or coronary artery bypass grafting (CABG)
* via median sternotomy

Exclusion Criteria:

* Surgery on an emergency basis (level 1 or 2, <2 hours)
* An ejection fraction <30%
* Patient on extracorporeal membrane oxygenator (ECMO),
* Presence of an intra-aortic balloon pump (IABP)
* Preoperative vasopressors or inotropes
* Severe pre-existing liver disease (Child B or C)
* Severe kidney disease (Glomerular filtration rate (GFR) <30 (mL/min/1·73m²))
* An allergy to ropivacaine
* Planned circulatory arrest
* BMI >35
* Weight <50 kg
* Opioid tolerant (oral morphine equivalent >60mg per day for >1 week prior to admission)
* Unable to provide valid consent to study prior to surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 1 month
  Number of patients recruited to the study
Adherence rate | Until measurement of quality of recovery at 72 hours
  The number of patients with no protocol violations
Primary outcome measurement rate (quality of recovery 15 index) | 72 hours
  The number of patients completing the quality of recovery 15 (QoR-15) index
Combined major block-related adverse event rate | Until block catheter is removed at 72 hours
  The number of patients experiencing a major block-related adverse event including pneumothorax, local anesthetic systemic toxicity (LAST) or allergic reaction.

SECONDARY OUTCOMES:
Quality of recovery 15 index (QoR-15) | 48, 72 hours
  The quality of recovery (QoR-15) questionnaire includes five domains of recovery after surgery: patient support, comfort, emotions, physical independence, and pain. Each item is graded on an eleven-point Likert scale with QoR-15 scores ranging from 0 (extremely poor quality of recovery) to 150 (excellent quality of recovery).
Pain scores | 24, 48, 72 hours
  Measured by numeric rating scale (NRS). The NRS has possible scores from 0 to 10 with higher numbers indicating worse pain.
Opioid use | 24, 48, 72 hours
  Measured by oral morphine equivalents (OME) in milligrams

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Bailey JG, Hendy A, Neira V, Chedrawy E, Uppal V. Continuous serratus anterior block for sternotomy analgesia after cardiac surgery: a single-centre feasibility study. Br J Anaesth. 2025 Apr;134(4):1161-1169. doi: 10.1016/j.bja.2024.11.042. Epub 2025 Jan 24. PMID 39863465